CLINICAL TRIAL: NCT05802563
Title: Pattern Recognition in Heart Rate Variability Using Fitness Trackers in Cardiovascular Disease
Brief Title: Machine Learning Enabled Time Series Analysis in Medicine
Acronym: ME-TIME
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: HagaZiekenhuis (Other)
Collaborators: Delft University of Technology (Other)
Responsible Party: Principal Investigator, Ivo van der Bilt, Principal Investigator, HagaZiekenhuis
Other Study IDs: metime
Record Dates: First submitted 2023-03-27; First posted 2023-04-06 (Actual); Last update posted 2023-04-07 (Actual); Status verified 2023-04

CONDITIONS: Atrial Fibrillation; Heart Failure, Systolic
Keywords: cardiovascular disease; Artificial intelligence; machine learning
MeSH Terms: conditions — Atrial Fibrillation; Heart Failure, Systolic; Cardiovascular Diseases | interventions — Fitness Trackers

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Heart Failure: Study participants with systolic heart failure (Left ventricular ejection fraction < 35%) without documented atrial fibrillation
  Interventions: Device: fitness tracker
- Atrial Fibrillation: Study participants with documented atrial fibrillation without heart failure
  Interventions: Device: fitness tracker
- Reference: Individuals without cardiovascular disease
  Interventions: Device: fitness tracker

INTERVENTIONS:
Device: fitness tracker — Study subjects will wear a Fitbit fitness tracker
  Other Names: Fitbit Charge 5, Fitbit Inspire 2

SUMMARY:
The goal of this observational cohort study is to investigate the potential of fitness trackers in combination with machine learning algorithms to identify cardiovascular disease specific patterns.

Two hundred participants will be enrolled:

1. 50 with heart failure
2. 50 with atrial fibrillation
3. 100 (healthy) individuals without the former two conditions

All participants are given a Fitbit device and monitored for three months. Researchers will compare differences in heart rate variability patterns between the groups and devise a machine learning algorithm to detect these patterns automatically.

ELIGIBILITY:
Inclusion Criteria:

* systolic heart failure (LVEF < 35%)
* Atrial fibrillation without heart failure
* Individuals without cardiovascular disease

Exclusion Criteria:

* > 85 years old
* Recent pulmonary venous antrum isolation procedure (<1 year)
* (end stage) kidney failure
* (end stage) liver failure
* Study participants with known systemic active inflammatory disease
* Study participants with impaired mental state
* Inability to use a fitness tracker or mobile phone
* Impaired cognition and inability to understand the study protocol

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All included participants will receive an electrocardiogram.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2022-05-24 (Actual); Primary Completion 2023-09-01 (Estimated); Study Completion 2023-09-01 (Estimated)

PRIMARY OUTCOMES:
Cardiovascular disease detection with an AI algorithm | Three months
  adequate sensitivity/specificity in an algorithm to detect atrial fibrillation and heart failure

SECONDARY OUTCOMES:
Detection of absence of cardiovascular disease | Three months

CONTACTS AND LOCATIONS:
Locations (1):
- HagaZiekenhuis, The Hague, South Holland, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
We are planning to release the full data set in the future.
Supporting Information: Study Protocol, Analytic Code
Time Frame: Expected release in 2026
Access Criteria: * Research institute
  * Open Access (full disclosure of results)
  * Clear data analysis plan